CLINICAL TRIAL: NCT00196833
Title: Prospective and Retrospective Register Study of the German Breast Group (GBG) for Diagnosis and Treatment of Breast Cancer in Pregnancy
Brief Title: Breast Cancer in Pregnancy Register Study
Acronym: BCP
Status: Recruiting | Type: Observational
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: Goethe University (Other)
Responsible Party: Sponsor
Other Study IDs: GBG 29; BIG 2-03 (Other: BIG)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer in Pregnancy; Prospective and Retrospective Register; Study
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Tumour and placenta specimens are collected
Oversight: Data Monitoring Committee: No

SUMMARY:
Women who were diagnosed with breast cancer during their pregnancy may be registered in this trial.

Data is collected on the foetal outcome 4 weeks after delivery, maternal outcome of pregnancy as well as the breast cancer therapy applied (treatment, response to chemotherapy, type of surgery), diagnostic procedures applied (palpation, US, mammogram) and the outcome of mother and child after 5 years of therapy.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer malignancy in women of childbearing age after the age of 25 years. Since the incidence of breast cancer under the age of 40 is increasing, and women tend to delay pregnancy into later reproductive years, the coincidence of pregnancy and breast cancer is increasing. About 1 in 1,000 pregnancies is complicated by breast cancer. Nevertheless, little is known about the right therapy for the mother and the unborn child. We are therefore carrying out a trial, collecting prospective and retrospective data about pregnant women, with histological confirmed breast cancer. Data on the biology of the tumour and placenta tissues is also collected. The anonymous data is collected in a database.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: Women with histologically confirmed breast cancer during pregnancy
* Cohort 2: Patients ≤ 40 years with histological confirmed breast cancer who are not pregnant (patients who have been pregnant recently can also be collected into this cohort)
* Informed consent for data collection (for prospective participants) and biomaterial collection. For retrospective participants an informed consent is not required as long as the data are anonymously captured

Exclusion Criteria:

* Cohort 1: Diagnosis of breast cancer outside the period of pregnancy
* Cohort 2: Age at diagnosis of breast cancer > 40 years

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cohort 1: Women with histologically confirmed breast cancer during pregnancy
  Cohort 2: Young women (age ≤ 40 years) with histologically confirmed breast cancer (outside of pregnancy or recently pregnant)
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2003-04; Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sibylle Loibl, Prof. Dr., Principal Investigator — GBG Forschungs GmbH
Locations (1):
- German Breast Group, Neu-Isenburg, Hesse, Germany

REFERENCES:
- [Derived] Loibl S, Han SN, von Minckwitz G, Bontenbal M, Ring A, Giermek J, Fehm T, Van Calsteren K, Linn SC, Schlehe B, Gziri MM, Westenend PJ, Muller V, Heyns L, Rack B, Van Calster B, Harbeck N, Lenhard M, Halaska MJ, Kaufmann M, Nekljudova V, Amant F. Treatment of breast cancer during pregnancy: an observational study. Lancet Oncol. 2012 Sep;13(9):887-96. doi: 10.1016/S1470-2045(12)70261-9. Epub 2012 Aug 16. PMID 22902483
- See also: Click here for more information about this study: Breast Cancer in Pregnancy — http://www.germanbreastgroup.de